CLINICAL TRIAL: NCT04403698
Title: The Use of Buffered Soluble Alendronate 70 mg (Steovess/Binosto) After Denosumab Discontinuation to Prevent Increase in Bone Turnover
Brief Title: The Use of Steovess/Binosto After Denosumab Discontinuation to Prevent Increase in Bone Turnover
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Amgen (Industry); EffRx Pharmaceuticals SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BC-6072
Record Dates: First submitted 2020-05-19; First posted 2020-05-27 (Actual); Results first posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-10

CONDITIONS: Erosive Osteoarthritis

STUDY DESIGN:
Intervention Model Description: 40 subjects randomized in 2 groups (n=20). 1 group will receive effervescent alendronate treatment for 24 weeks, the other group will receive the same treatment for 48 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 24 weeks (Experimental): Subject receiving alendronate treatment for 24 weeks (n = 20)
  Interventions: Drug: Alendronate Effervescent Oral Tablet
- 48 weeks (Experimental): Subject receiving alendronate treatment for 48 weeks (n = 20)
  Interventions: Drug: Alendronate Effervescent Oral Tablet

INTERVENTIONS:
Drug: Alendronate Effervescent Oral Tablet — At the earliest three months but no later than four months after the last denosumab injection, subjects will be randomized to effervescent alendronate administered for either 24 or 48 weeks

SUMMARY:
It is hypothesized that effervescent alendronate will be able to maintain bone turnover markers within the pre-menopausal reference range and thereby reducing the likelihood of bone turnover associated changes (rebound effect), after discontinuation of denosumab treatment in a non-osteoporotic population.

DETAILED DESCRIPTION:
Denosumab discontinuation is associated with a rebound effect in bone turnover and loss in bone mass density. These changes resulted in an increase of fracture incidence in patients with postmenopausal osteoporosis back to background levels. However, no excess in fracture incidence was observed. Amongst patients who presented with vertebral fractures after treatment discontinuation, there was a slightly higher incidence of multiple vertebral fractures in patients discontinuing Prolia versus those who discontinued the placebo treatment.

A 2 year, randomized, crossover study demonstrated that alendronate intake after discontinuing denosumab treatment, lead to remaining stable bone mass densitometry (BMD) values in postmenopausal women.

In a study within a non-osteoporotic study population, ongoing at our department, increases in bone turnover are to be expected as soon as patients end study participation (i.e. open label treatment with denosumab, Prolia, anti-RANK ligand inhibition).

It is currently recommended that alternative anti-resorptive therapy may be warranted after Prolia discontinuation. One study describes the use of oral alendronate after denosumab therapy to maintain bone mineral density. However, gastro-intestinal upset and tolerability, as well as difficulty in swallowing pills may limit oral alendronate compliance. To attenuate this concern, buffered soluble (effervescent) alendronate 70 mg, developed with the aim to improve the gastrointestinal tolerability through full dissolution of alendronate in buffered palatable solution before ingestion, will be used.

This study wants to provide a follow up and study wether the use of effervescent alendronate after previous denosumab treatment can prevent a rebound effect in bone turnover that is to be expected when denosumab is discontinued. Subjects that completed our erosive hand osteoarthritis (OA) study and therefore discontinued denosumab 60 mg/every 3 months, will receive alendronate. Moreover, the study wants to asses if there is difference between using alendronate for six or twelve months, starting at the earliest three months but no later than four months after the last injection of denosumab.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have completed the 48 weeks of the randomised placebo-controlled study phase followed by the 96 weeks open label denosumab 60 mg SC every 3 months phase. (EudraCT number: 2015-003223-53)
* Last denosumab injection minimal 3 months or maximum 4 months before baseline
* Able and willing to give written informed consent and to comply with the requirements of the study protocol

Exclusion Criteria:

* Patients with clinically significant hypersensitivity to any of the components of effervescent alendronate.
* Patient who is pregnant or planning pregnancy
* Female subjects who are breast-feeding.
* History of osteonecrosis of the jaw, and/or recent (within 3 months) tooth extraction or other unhealed dental surgery; or planned invasive dental work during the study
* Subject has any kind of disorder that compromises the ability of the subject to give written informed consent and/or to comply with study procedures
* Hypocalcaemia.
* Oesophageal disease, gastritis, duodenitis, ulcers, or with a recent history (within the previous year) of major gastro-intestinal disease such as peptic ulcer, or active gastro-intestinal bleeding, or surgery of the upper gastro-intestinal tract other than pyloroplasty.
* Abnormalities of the oesophagus and other factors which delay oesophageal emptying such as stricture or achalasia.
* Inability to stand or sit upright for at least 30 minutes.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2022-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Wittoek, Prof. dr., Principal Investigator — Ghent Universitary Hospital
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD that underlie results in a publication will be shared
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months after publication. Data will stay available for 3 years after publication
Access Criteria: acces will be provided upon reasonable request from researchers with a sound clinical research question

REFERENCES:
- [Background] Miller PD, Bolognese MA, Lewiecki EM, McClung MR, Ding B, Austin M, Liu Y, San Martin J. Effect of denosumab on bone density and turnover in postmenopausal women with low bone mass after long-term continued, discontinued, and restarting of therapy: a randomized blinded phase 2 clinical trial. Bone. 2008 Aug;43(2):222-229. doi: 10.1016/j.bone.2008.04.007. Epub 2008 Apr 26. PMID 18539106
- [Background] Brown JP, Roux C, Torring O, Ho PR, Beck Jensen JE, Gilchrist N, Recknor C, Austin M, Wang A, Grauer A, Wagman RB. Discontinuation of denosumab and associated fracture incidence: analysis from the Fracture Reduction Evaluation of Denosumab in Osteoporosis Every 6 Months (FREEDOM) trial. J Bone Miner Res. 2013 Apr;28(4):746-52. doi: 10.1002/jbmr.1808. PMID 23109251
- [Background] Cummings SR, Ferrari S, Eastell R, Gilchrist N, Jensen JB, McClung M, Roux C, Torring O, Valter I, Wang AT, Brown JP. Vertebral Fractures After Discontinuation of Denosumab: A Post Hoc Analysis of the Randomized Placebo-Controlled FREEDOM Trial and Its Extension. J Bone Miner Res. 2018 Feb;33(2):190-198. doi: 10.1002/jbmr.3337. Epub 2017 Nov 22. PMID 29105841
- [Background] Freemantle N, Satram-Hoang S, Tang ET, Kaur P, Macarios D, Siddhanti S, Borenstein J, Kendler DL; DAPS Investigators. Final results of the DAPS (Denosumab Adherence Preference Satisfaction) study: a 24-month, randomized, crossover comparison with alendronate in postmenopausal women. Osteoporos Int. 2012 Jan;23(1):317-26. doi: 10.1007/s00198-011-1780-1. Epub 2011 Sep 17. PMID 21927922
- [Background] Hodges LA, Connolly SM, Winter J, Schmidt T, Stevens HN, Hayward M, Wilson CG. Modulation of gastric pH by a buffered soluble effervescent formulation: A possible means of improving gastric tolerability of alendronate. Int J Pharm. 2012 Aug 1;432(1-2):57-62. doi: 10.1016/j.ijpharm.2012.04.073. Epub 2012 May 4. PMID 22564778

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Alendronate 70 mg Weekly for 24 Weeks: Subject receiving alendronate treatment for 24 weeks (n = 15)
  Alendronate Effervescent Oral Tablet: At the earliest three months but no later than four months after the last denosumab injection, subjects were randomized to effervescent alendronate administered for 24 weeks
- Treatment Alendronate 70 mg Weekly for 48 Weeks: Subject receiving alendronate treatment for 48 weeks (n = 15)
  Alendronate Effervescent Oral Tablet: At the earliest three months but no later than four months after the last denosumab injection, subjects will be randomized to effervescent alendronate administered for 48 weeks
Period: Overall Study
Arm/Group | Treatment Alendronate 70 mg Weekly for 24 Weeks | Treatment Alendronate 70 mg Weekly for 48 Weeks
Started | 15 | 15
Completed | 13 | 13
Not Completed | 2 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Alendronate 70 mg Weekly for 24 Weeks | Treatment Alendronate 70 mg Weekly for 48 Weeks | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (7.7) | 64.7 (8.9) | 64.0 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 3 | 4 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 15 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
mean treatment duration with denosumab (days) [Mean (Standard Deviation); unit: days] | 813 (165) | 751 (174) | 782 (170)
mean time since last denosumab injection (days) [Mean (Standard Deviation); unit: days] | 89 (7) | 94 (8) | 91 (8)
N-terminal propeptide of type I procollagen (PINP) [Mean (Standard Deviation); unit: microgram/L] | 10.15 (5.5) | 8.97 (10.6) | 9.56 (8.3)
C-terminal telopeptide of type I collagen (CTX-I) [Mean (Standard Deviation); unit: ng/ml] | 0.057 (0.03) | 0.071 (0.06) | 0.064 (0.05)
Bone mineral density hip [Mean (Standard Deviation); unit: g/cm2] | 0.85 (0.10) | 0.80 (0.08) | 0.83 (0.11)
Bone mineral density spine [Mean (Standard Deviation); unit: g/cm2] | 1.16 (0.11) | 1.11 (0.16) | 1.14 (0.13)

OUTCOME MEASURES:

1. Primary Outcome: CTX-I (C-terminal Telopeptide of Type I Collagen ) Bone Turnover Marker Levels
Description: Difference in bone turnover marker C-terminal telopeptide of type I collagen (CTX-I) after 48 weeks. Comparisons made within and between both treatment arms
Time Frame: 48 weeks
Measure: Geometric Mean (Standard Error); unit: ng/ml
Groups:
- 24 Weeks: Subject receiving alendronate treatment for 24 weeks (n = 15)
- 48 Weeks: Subject receiving alendronate treatment for 48 weeks (n = 15)
Arm/Group | 24 Weeks | 48 Weeks
Number analyzed (Participants) | 15 | 15
ng/ml
  Baseline | 0.05 (0.06) | 0.06 (0.06)
  Week 48 | 0.63 (0.33) | 0.33 (0.33)
Statistical Analysis 1: Comparison: 24 Weeks vs 48 Weeks; linear mixed models were used to compare bone turnover markers (CTX-I) between both treatment groups. These models were performed with an intention to treat approach, where drop-outs were considered as non-responders. The models accounted for repeated measures; Test type: Superiority; p < 0.01, Mixed Models Analysis

2. Primary Outcome: PINP (N-terminal Propeptide of Type I Procollagen) Bone Turnover Marker Levels
Description: Difference in Bone Turnover Marker N-terminal propeptide of type I procollagen (PINP) After 48 Weeks. Comparisons are made both within and between both treatment arms.
Time Frame: 48 weeks
Measure: Geometric Mean (Standard Error); unit: microgram/L
Arm/Group | 24 Weeks | 48 Weeks
Number analyzed (Participants) | 15 | 15
microgram/L
  Baseline | 8.1 (0.41) | 4.6 (0.41)
  Week 48 | 78.9 (0.44) | 39.5 (0.44)
Statistical Analysis 1: Comparison: 24 Weeks vs 48 Weeks; linear mixed models were used to compare bone turnover markers (PINP) between both treatment groups. These models were performed with an intention to treat approach, where drop-outs were considered as non-responders. The models accounted for repeated measures; Test type: Superiority; p = 0.05, Mixed Models Analysis

3. Secondary Outcome: Number of Patients With CTX-I (C-terminal Telopeptide of Type I Collagen )Levels Above the Reference Range at Week 48
Description: The number of patients that do not maintain C-terminal telopeptide of type I collagen (CTx-I) levels within the bone turnover marker reference range at week 48.
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Treatment Alendronate 70 mg Weekly for 24 Weeks: Subject receiving alendronate treatment for 24 weeks (n = 15)
- Treatment Alendronate 70 mg Weekly for 48 Weeks: Subject receiving alendronate treatment for 48 weeks (n = 15)
Arm/Group | Treatment Alendronate 70 mg Weekly for 24 Weeks | Treatment Alendronate 70 mg Weekly for 48 Weeks
Number analyzed (Participants) | 15 | 15
Participants | 5 | 0
Statistical Analysis 1: Comparison: Treatment Alendronate 70 mg Weekly for 24 Weeks vs Treatment Alendronate 70 mg Weekly for 48 Weeks; A Fisher's exact test was used to assess differences in patient numbers exceeding reference ranges between both treatment groups at week 48; Test type: Superiority; p = 0.042, Fisher Exact

4. Secondary Outcome: The Number of Patients PINP (N-terminal Propeptide of Type I Procollagen) Above Reference Range at Week 48
Description: The number of patients that do not maintain N-terminal propeptide of type I procollagen (PINP) levels within the bone turnover marker reference range at week 48
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Alendronate 70 mg Weekly for 24 Weeks | Treatment Alendronate 70 mg Weekly for 48 Weeks
Number analyzed (Participants) | 15 | 15
Participants | 5 | 0
Statistical Analysis 1: Comparison: Treatment Alendronate 70 mg Weekly for 24 Weeks vs Treatment Alendronate 70 mg Weekly for 48 Weeks; A Fisher's exact test was used to assess differences in patient numbers exceeding reference ranges between both treatment groups; Test type: Superiority; p = 0.042, Fisher Exact

5. Secondary Outcome: Bone Mass Density at the Spine After 48 Weeks
Description: Difference in bone mass density at the spine after 48 Weeks. Comparisons are made both within and between both treatment arms
Time Frame: 48 weeks
Measure: Geometric Mean (Standard Error); unit: g/cm2
Arm/Group | Treatment Alendronate 70 mg Weekly for 24 Weeks | Treatment Alendronate 70 mg Weekly for 48 Weeks
Number analyzed (Participants) | 15 | 15
g/cm2
  Baseline | 1.16 (0.03) | 1.11 (0.03)
  Week 48 | 1.10 (0.03) | 1.11 (0.03)

6. Secondary Outcome: Bone Mass Density at the Hip After 48 Weeks
Description: Difference in Bone Mass Density at the hip After 48 Weeks. Comparisons are made both within and between both treatment arms.
Time Frame: 48 weeks
Measure: Geometric Mean (Standard Error); unit: g/cm2
Arm/Group | Treatment Alendronate 70 mg Weekly for 24 Weeks | Treatment Alendronate 70 mg Weekly for 48 Weeks
Number analyzed (Participants) | 15 | 15
g/cm2
  Baseline | 0.85 (0.03) | 0.80 (0.03)
  Week 48 | 0.85 (0.03) | 0.81 (0.03)

ADVERSE EVENTS:
Time Frame: Adverse events data was collected during the 48 weeks of the trial duration.
Groups:
- Alendronate 24 Weeks: Subject receiving alendronate treatment for 24 weeks and daily oral supplements of calcium and vitamin D for 48 weeks (n = 15)
- Alendronate 48 Weeks: Subject receiving alendronate treatment for 48 weeks daily oral supplements of calcium and vitamin D (n = 15)
Arm/Group | Alendronate 24 Weeks | Alendronate 48 Weeks
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 1/15 | 0/15
Other Adverse Events (participants affected / at risk) | 10/15 | 12/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alendronate 24 Weeks (N=15) | Alendronate 48 Weeks (N=15)
Colonic ulcers (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alendronate 24 Weeks (N=15) | Alendronate 48 Weeks (N=15)
Arterial hypertension (Cardiac disorders) | 1 (1) | 1 (1)
Infections (Infections and infestations) | 3 (3) | 4 (7) — Infections (mostly being upper airway infections)
stomach and stool problems (Gastrointestinal disorders) | 5 (9) | 6 (8) — Gastro-intestinal adverse events including stomach pain, diarrhoa, loss of appetite, nausea,..
muscular pain and joint pain (Musculoskeletal and connective tissue disorders) | 4 (6) | 5 (8)
Headache and dizziness (Nervous system disorders) | 3 (3) | 1 (1)
Cough (non-infectious) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Itch (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Throat pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Blurry vision and eye dryness (Eye disorders) | 1 (1) | 2 (2)
General malaise (General disorders) | 0 (0) | 1 (1)
Bone fractures (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0)
Hypercholesterolemia (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Hair loss (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The target number of participants was not reached and therefore underpowered. The study should be repeated on a higher number of participants and with a longer follow-up time to estimate clinical consequences on long term.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-08-09): https://cdn.clinicaltrials.gov/large-docs/98/NCT04403698/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-04): https://cdn.clinicaltrials.gov/large-docs/98/NCT04403698/SAP_001.pdf